CLINICAL TRIAL: NCT07259785
Title: Comparison of the Effects of Serratus Posterior Superior Intercostal Plane Block Versus Costoclavicular Brachial Plexus Block on Postoperative Pain and Hemidiaphragmatic Paralysis in Arthroscopic Shoulder Surgeries
Brief Title: SPSIPB vs CCB in Arthroscopic Shoulder Surgeries
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Oguz Gundogdu, Associate Professor, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-10/12
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain; Shoulder Arthoscopy
Keywords: postoperative pain; shoulder arthroscopy; regional anesthesia; costoclavicular brachial plexus block; serratus posterior superior intercostal plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPSIPB (Active Comparator): SPSIPB will be performed on the ipsilateral side of the patient right after the anesthesia induction with the patients in lateral position.The ultrasound probe was placed 2-3 cm medial to the scapular spine to visualize the trapezius, rhomboid major, and serratus posterior superior muscles. At the level of the 2nd-3rd ribs, a needle was advanced into the plane between the serratus posterior superior muscle and the ribs. After confirming the placement of the needle tip with negative aspiration, 30 mL of 0.25% bupivacaine was injected. The block was performed unilaterally, targeting the shoulder undergoing surgery.
  Interventions: Procedure: Serratus posterior superior intercostal plane block
- CCBPB (Active Comparator): CCBPB will be performed on the ipsilateral side of the patient right after the anesthesia induction with the patients in supine position. For CCBPB, a high frequency linear transducer of the USG is placed in the medial infraclavicular fossa parallel and next to the clavicle to identify the axillary artery. The transducer is then tilted cephalad to image the brachial plexus and the artery in a perpendicular orientation between the subclavius muscle and the serratus anterior. The needle is advanced in-plane in a lateral-to-medial direction, adjusting the angle to reach the space in between the three cords. 15 mL of 0.25% bupivacaine is administered.
  Interventions: Procedure: Costoclavicular brachial plexus block

INTERVENTIONS:
Procedure: Serratus posterior superior intercostal plane block — 30 mL of 0.25% bupivacaine
  Arms: SPSIPB
Procedure: Costoclavicular brachial plexus block — 15 mL of 0.25% bupivacaine
  Arms: CCBPB

SUMMARY:
The aim is to compare the postoperative analgesic and hemidiaphragmatic effects of Serratus Posterior Superior Intercostal Plane Block (SPSIPB) versus CostoClavicular Brachial Plexus Block (CCBPB) in patients undergoing arthroscopic shoulder surgery.

DETAILED DESCRIPTION:
Patients were divided into two randomized groups: Group 1 (SPSIPB group, n=15) and Group 2 (CCBPB group, n=15). All patients will receive the same standard general anesthesia per hospital protocol. All blocks will be applied with the same ultrasonography and block equipment, and by the same physician. Before the anesthesia induction, ipsilateral diaphragmatic excursion will be measured via Ultrasonography (USG). After the anesthesia induction, patients in Group 1 will receive Serratus Posterior Superior Intercostal Plane Block (SPSIPB) with 30 mL of 0.25% bupivacaine. Patients in Group 2 will receive Costoclavicular Brachial Plexus Block (CCBPB) with 15 mL of 0.25% bupivacaine. All patients will receive Paracetamol 1gr and Dexketoprofen 50mg intravenous (IV) 10 minutes prior to skin closure. After 30 minutes of emergence from anesthesia (upon reaching 9 points on modified Aldrete scoring), ipsilateral diaphragmatic excursion will be assessed again. Pre- and postblock excursion differences will be recorded. Routine analgesic procedure consisting of 3x1gr Paracetamol IV and 2x50mg Dexketoprofen IV will be followed postoperatively for 24 hours. Numeric Rating Scale (NRS) will be used to assess postoperative pain on 1st, 6th, 12th, 18th and 24th hours after the surgery. Quality of Recovery-15 Patient Survey will be done both preoperatively for a baseline score, and postoperatively at 24th hour to assess the quality of recovery from the patients' view. Tramadol 50mg IV will be administered as a rescue analgesic for all patients if NRS score is equal to or higher than 4. Total Tramadol consumption will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years of age who underwent unilateral elective arthroscopic shoulder surgery under general anesthesia and were American Society of Anesthesiologists (ASA) score I-II-III according to the ASA risk classification.

Exclusion Criteria:

* patients who did not give consent,
* patients with coagulopathy,
* patients with signs of infection at the block application site,
* patients using anticoagulants,
* patients with local anesthetic drug allergies,
* patients with unstable hemodynamics,
* patients who could not cooperate during postoperative pain assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) Scores | Postoperative 24 hours
  Numerical rating scale is used for pain assessment. The scores of the numerical rating scale changes between 0 to 10 points. 10 points mean "the most severe pain that the patient ever had". 0 point means "there is no pain." Higher scores mean worse outcome.
Diaphragmatic Excursion Difference | Preoperatively right before the anesthesia induction, and postoperatively after 30 minutes of emergence from anesthesia (upon reaching 9 points on modified Aldrete scoring)
  Ipsilateral diaphragmatic excursions will be measured both preoperatively right before the anesthesia induction, and postoperatively after 30 minutes of emergence from anesthesia (upon reaching 9 points on modified Aldrete scoring). A diaphragmatic excursion change of up to 25% indicates no nerve involvement, a change between 25%-75% indicates partial involvement, and a change exceeding 75% indicates complete involvement of the phrenic nerve.

SECONDARY OUTCOMES:
Total tramadol consumption | Postoperative 24 hours
  Postoperative total opioid need was recorded as "milligram" in unit.
Quality of Recovery-15 Patient Survey (QoR-15) | Preoperatively and Postoperatively at 24th hour
  The widespread use of minimally invasive interventions to reduce postoperative mortality and morbidity, combined with the implementation of Enhanced Recovery After Surgery (ERAS) protocols, has heightened overall interest in the postoperative recovery period and the importance of outcome evaluation. To address the emerging needs in this field, new tools prioritizing patient satisfaction have been developed alongside traditional scales that measure classical parameters. The Quality of Recovery-15 Patient Survey (QoR-15) stands out as one of the most up-to-date and reliable examples among these tools. The survey is done both preoperatively to record patients' baseline score, and postoperatively at 24th hour. Higher scores mean better quality of recovery after surgery. Mininum and maximum scores can be '0 (zero)' and '150 (one hundred and fifty)' respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Oğuz Gündoğdu, Principal Investigator — Sivas Cumhuriyet University School of Medicine, Anesthesiology and Reanimation
Locations (1):
- Sivas Cumhuriyet University, Sivas, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No